CLINICAL TRIAL: NCT01671553
Title: Helping Smokers to Quit Via the Smoke-free Teen Contest 2011: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Sophia Siu-chee Chan, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COSH-SmokefreeTeen
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Comparative Effectiveness Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling group (Experimental): Study participants in the intervention group were received an intensive smoking cessation telephone counselling with 2-weeks free and 6-weeks discount nicotine replacement therapy (NRT).
  Interventions: Behavioral: Counseling group
- Control group (No Intervention): Study participants in the control group were not received any quitting assistance other than the self-help materials provided by Hong Kong Council on Smoking and Health (COSH).

INTERVENTIONS:
Behavioral: Counseling group — The content for the brief counseling group adopts a AWARD approach including asking the smoking habit, warning about the health risks associated with smoking, advising the smokers to quit, referring to specialized service, and repeating the above message. Additional telephone follow-up counseling at 1, 2, 3 and 8-week will be made to the participants in this group.
  Arms: Counseling group

SUMMARY:
Background The home is the primary source of SHS exposure. The scientific evidence shows that there is no risk-free level of exposure to SHS that stop smoking is the sole way to completely eliminate the risk of SHS exposure. Although research studies indicated that smoking bans in restaurants, bars, and workplaces can significantly reduce the level of SHS exposure, governments lack the authority to restrict smoking in homes. Therefore, parental cessation is a more effective means to reduce the SHS exposure.

Aim The aims are (1) to promote smoking cessation in the community and (2) assess the effect of different smoking cessation approaches through the Smoke-free Teen Contest. The specific objectives of the study are to test the effectiveness of different smoking cessation approaches on quit rate and change in smoking behaviours among smokers who are referred by Hong Kong Council on Smoking and Health (COSH).

Methods The referred smokers were nominated by primary 1 to secondary 3 students who joined the Smoke-free Teen Contest organized by COSH. Two domains of outcome will be assessed: (1) the primary outcome is the self-reported 7-day point prevalence (pp) quit rate at 6 months and (2)the secondary outcomes included (i) biochemical validated quit rate at 6 months and (ii) rate of smoking reduction by at least of half and (iii) number of quit attempts at 6 months.

Procedure Smokers, who are referred by the Hong Kong Council on Smoking and Health (COSH), were nominated by primary 1 to secondary 3 students joined Smoke-free Teen Contest organized by COSH. Those smokers will be randomized into two groups (Intervention group and Control group) using the clustered randomization method by school. After the clustered randomization, the oral consent of eligible subjects were obtained to the study through telephone interview. Intervention group will receive 1,2,3, 8-week and 6-month telephone follow-up after baseline, while control group will only receive 6-month telephone follow-up after baseline. Those participants who reported to have stopped smoking will be invited for biochemical validation of smoking status at 6-month follow-up.

Hypothesis We hypothesize that the intensive telephone counselling plus NRT treatment will lead to significant increases in rates of smoking cessation in the intervention groups than the control group.

DETAILED DESCRIPTION:
Smoking is the single most preventable cause of deaths in Hong Kong and the smoking prevalence was about 11.8% (20.5% in males and 3.6% in females) in 2008. It was estimated that smoking accounts for about one fifth of all deaths and kills about 5,700 people per year. Smoking has been associated with serious damage to health at all ages, leading to cancers, heart diseases, stroke, chronic lung diseases, and many other health problems. It was estimated in 1998 that a total of US$688 million medical cost were attributed to smoking-related diseases annually, with active smoking accounted for 77% and passive smoking 23% of the total cost. However, it is difficult for smokers to quit smoking without assistance because smoking is addictive, and most smokers prefer to try and quit on their own rather than seeking treatment, thus it is hard to reach those smokers who do not present themselves for treatment. On the other hand, a previous study also indicated that high quit rate (38%) could be achieved for those smokers who received a 6-week supply of free NRT plus telephone counselling and self-help materials.

Consistent findings from previous studies demonstrated that social support appears to be one of the strongest determinants of success at quitting smoking and remaining abstinent. Ward and Klesges showed that social (family) support affects smoking outcome and may influence readiness to quit. In a US study, family support was reported to be the most significant predictor, compared to peer and significant-other support, on the experiential and behavioral processes of change in a smoking cessation program for adult smokers. Similar results were also found in a local study on the motivation to reduce smoking among smokers who are not willing to quit. It is therefore imperative to involve a family member as the first point of contact in the health care system regarding supporting their smoking family members in the quitting process.

In Hong Kong, 33.6% of fathers and 2.6% of mothers smoke. Nevertheless, only 1.8% male smokers had tried smoking cessation service and among those who had not tried any, 86.1% reported that they would not try the service. Establishing rapport with schools and building capacity in tobacco control in students could be a feasible way to engage smokers in tobacco control advocacy. This could also help smokers who may not have access to services which assists them in quitting smoking.

To fill those aforementioned gaps, in this proposed project, all primary school students and junior forms of secondary school students are mobilized for the establishment of smoke-free homes. They play an active role in advocating for a 'Smoke-free Environment' in their home by nominating, encouraging and supporting their family members and relatives to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Able to communicate in Cantonese
* Intend to quit smoking

Exclusion Criteria:

* Smokers who are psychologically or physically unable to communicate
* Currently following other forms of smoking cessation programme
* Have a previous history of allergy to NRT patch or gum

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The self-reported 7-day point prevalence (pp) quit rate at 6 months | Six months
  Whether the participant has quitted smoking in the past seven days at the time point of 6 months

SECONDARY OUTCOMES:
Biochemical validated quit rate at 6 months | Six months
  * Test the cotinine level in the saliva provided by the participants
  * Rate of smoking reduction by at least of half
  * Number of quit attempts at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophia SC Chan, PhD, Principal Investigator — HKU
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China